CLINICAL TRIAL: NCT00797199
Title: Short-term Evaluations of Breast Tissue Change in Post-menopausal Women Using Optical Breast Spectroscopy (OBS)
Brief Title: Monitoring of Breast Tissue Change Due to Hormone Replacement Therapy in Post-menopausal Women Using OBS
Acronym: TiBS-HRT
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: TiBS-HRT
Record Dates: First submitted 2008-06-02; First posted 2008-11-25 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer Risk; Hormone Replacement Therapy; Optical Transillumination Spectroscopy; Optical Breast Spectroscopy; Transillumination Breast Spectroscopy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1-Treatment Group 1: Women receiving HRT treatment of Premarin.
- 2-Treatment Group 2: Women receiving combination HRT treatment of Premarin + Provera.
- 3- Treatment Group 3: Women receiving combination HRT treatment of Premarin + Prometrium.
- 4- Controls: Women not on HRT or healthy controls.

SUMMARY:
Hormone Replacement Therapy (HRT) is a double edged sword: it can alleviate the effects of menopause for a significant proportion of the female population, however for a smaller proportion, it will induce a significant increase in their short-term and lifetime risk to develop breast cancer (BC). Fewer women are prescribed HRT compared to a decade ago due to concerns pertaining to BC by both physicians and patients. By developing a technology that could identify women at risk for the adverse effects of HRT, during the first few months of its use, physicians may offer HRT to a wider proportion of the female population during menopause. More importantly, as it relates to BC prevention, such a technology will identify women at risk and provide a useful decision making tool regarding their care during the menopausal years.

DETAILED DESCRIPTION:
Hormone Replacement Therapy (HRT) provides many benefits to post-menopausal women, which have been overshadowed by an increase in breast cancer in women following HRT, resulting in a negative HRT cost-benefit ratio. Epidemiological studies show evidence of a direct association between HRT use and breast cancer incidence. This increase in incidence was also reflected in an increase of the mammographic breast density (MBD). Endogenous MBD is a well established risk factor for breast cancer which provides a high odds ratio (OR 4 - 6) towards breast cancer. Increases in MBD have been reported in women who initiate HRT, which is of concern as it potentially indicates a greater adverse effect of HRT on those individuals. In these cases, the majority of the incremental MBD increase manifests itself during the first year of use and decreases in the case of therapy cessation. The ability to detect changes in MBD in women commencing HRT treatment, without the ionizing radiation dose penalty imparted by mammography, thus permitting improved monitoring of MBD changes de to HRT, would certainly impact the debate on the applicability of HRT. Women identified as having increased MBD induced by HRT should discontinue its use or modify the prescription as increases in MBD potentially indicates an adverse ratio; women whose MBD has not been adversely affected by HRT can continue its use and reap the benefits of HRT (e.g. relief of climacteric symptoms, beneficial effects against osteoporosis and coronary heart disease).

Optical Breast Spectroscopy (OBS) is a safe and non-invasive optical technique that provides information on breast tissue composition and physiology state. Comparison of breast tissue status over time will provide information on changes in the MBD and breast cancer risk due to interventions such as HRT. To demonstrate that breast tissue status changes with HRT use, we will exploit existing algorithms correlating OBS with various biological outcomes. A completed study on a cohort of 300 healthy women (age 38 to 72) showed a high correlation between OBS optical parameters and Cumulus derived MBD. An ongoing study, to be completed Q3 2008 with an interim analysis available, suggests that OBS parameters can optically detect differences between the contralateral breasts of women with a unilateral carcinoma or ductal carcinoma in situ (DCIS) and healthy controls. Through these studies, two OBS algorithms ("density" and "risk") are available for application in the proposed study. The algorithms take OBS optical data as input and output OBS-derived percent breast density (PBD) and OBS-derived risk values. The aim of the study is to examine changes in OBS-derived PBD and OBS-derived risk values due to the initiation, use and cessation of HRT over a 1 year period. The case group will comprise a population of post-menopausal women who have elected to undergo a HRT regiment designed to last at least 1 year but had no prior HRT treatment. The comparison group (control) will comprise of post-menopausal women not on HRT and had no prior HRT treatment. OBS measurements will be assessed at intervals corresponding to: baseline (pre-HRT), 1 month, 3 months, 6 months, and 1 year after initiation of HRT use, and 3 months after cessation of treatment (in cases where HRT is discontinued within one year). Blood will be collected at baseline and at 3 months during treatment to examine changes in circulating hormones (estrogen, progesterone). Mammography will be performed at three months during treatment and compared to a screening mammogram (taken within a year prior to HRT treatment) to determine changes in breast density. A Papanicolaou test (or PAP smear) will be performed at baseline to assess endometrial changes. Changes in OBS derived PBD and MBD as well as other pertinent risk values will be examined as a function of time.

Four model groups will be monitored consisting of cases receiving treatments of Premarin, Premarin + Provera combination, or Premarin + Prometrium combination and controls not on HRT. A total of 20 women will be recruited into each group of the four groups. While the total number of women intended for recruitment is small, they are sufficient to enable us to demonstrate that OBS changes as function of MBD changes. Of further interest, we want to determine whether OBS can detect changes prior to changes to MBD in standard clinical setting. In particular, we aim to determine the magnitude of the effect size and the variance within the study groups for later initiation of a larger definitive clinical monitoring trail of HRT effects by OBS.

The long term clinical goal is the identification of women adversely affected by HRT by OBS as they can be advised of alternative methods with possible lower risk to benefit ratio to relieve climacteric symptoms. An overall effect will be a reduction in the population-based incidence of breast cancer while not withholding the beneficial effects of HRT to the majority of women during menopause.

ELIGIBILITY:
Cases

Inclusion Criteria:

* Post-menopausal
* Attending the Endocrinology clinic at SMH
* Will start HRT treatment

Exclusion Criteria:

* Current or Past HRT treatment
* Prior breast cancer
* Benign breast disease
* Bilateral breast biopsy
* Fine needle aspiration (FNA) within a year
* Cosmetic alteration (reduction/augmentation)
* Gynecological surgery
* Past or current chemo- therapeutic or prevention treatment

Controls

Inclusion Criteria:

* Not on HRT treatment

Exclusion Criteria:

* Current or Past HRT treatment
* Prior breast cancer
* Benign breast disease
* Bilateral breast biopsy
* Fine needle aspiration (FNA) within a year
* Cosmetic alteration (reduction/augmentation)
* Gynecological surgery
* Past or current chemo- therapeutic or prevention treatment

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Post-menopausal women attending the Endocrinology Clinic at St. Michael's Hospital (Toronto, Ontario, Canada) who have elected to undergo a 1-year HRT regiment but had no prior HRT treatment. The comparison group (control) will comprise of post-menopausal women not on HRT and had no prior HRT treatment. Controls will be recruited among women at the University Health Network or attending the Endocrinology Clinic at St. Michael's Hospital (Toronto, Ontario, Canada).
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2011-09; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Changes in OBS parameters | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Lothar Lilge, PhD, Principal Investigator — Ontario Cancer Institute, University Health Network, Toronto, Ontario, Canada M5G 2M9; Department of Biophysics and Bioimaging, University of Toronto, Toronto, Ontario, Canada M5G 2M9
Locations (2):
- Canada (2):
  - Princess Margaret Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario

REFERENCES:
- [Background] Blyschak K, Simick M, Jong R, Lilge L. Classification of breast tissue density by optical transillumination spectroscopy: optical and physiological effects governing predictive value. Med Phys. 2004 Jun;31(6):1398-414. doi: 10.1118/1.1738191. PMID 15259643
- [Background] Simick MK, Jong R, Wilson B, Lilge L. Non-ionizing near-infrared radiation transillumination spectroscopy for breast tissue density and assessment of breast cancer risk. J Biomed Opt. 2004 Jul-Aug;9(4):794-803. doi: 10.1117/1.1758269. PMID 15250768
- [Background] Blackmore KM, Knight JA, Jong R, Lilge L. Assessing breast tissue density by transillumination breast spectroscopy (TIBS): an intermediate indicator of cancer risk. Br J Radiol. 2007 Jul;80(955):545-56. doi: 10.1259/bjr/26858614. Epub 2007 May 30. PMID 17537757
- [Background] Simick MK, Lilge L. Optical transillumination spectroscopy to quantify parenchymal tissue density: an indicator for breast cancer risk. Br J Radiol. 2005 Nov;78(935):1009-17. doi: 10.1259/bjr/14696165. PMID 16249602